CLINICAL TRIAL: NCT06146244
Title: Comparison Between Value of Resonance Frequency Analysis (ISQ) in Implants Placed in Antral Area on Native Bone vs Value Obtained in Implants Placed in Antral Area on Regenerated Bone and Its Evolution After 3 Months
Brief Title: Comparison of ISQ in Implants Placed in Antral Area on Native Bone vs Regenerated Bone
Status: Completed | Type: Observational
Sponsor: European University of Madrid (Other)
Responsible Party: Principal Investigator, Barbara Molina Ponte, ASSOCIATE PROFESSOR, European University of Madrid
Other Study IDs: CIPI/18/008
Record Dates: First submitted 2023-11-14; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Implant Site Reaction
Keywords: Implant placement; native bone; regenerated bone; resonance frequency analysis; ISQ value; Ostell
MeSH Terms: interventions — Resonance Frequency Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — we performed an ostell mesuarement on dental implants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Native bone: the evolution of the SSI and its change after 3 months of placing the implant in native bone in the antral area
  Interventions: Device: resonance frequency analysis
- Regenerated Bone: the evolution of the SSI and its change after 3 months of placing the implant in regenerated bone in the antral area
  Interventions: Procedure: sinus lift; Device: resonance frequency analysis

INTERVENTIONS:
Procedure: sinus lift — Implant placement on grafted sinus vs antral autogenous bone
  Other Names: alveolar preservation
  Groups: Regenerated Bone
Device: resonance frequency analysis — analysis of the ISQ evolution and its changes after 3 months of placing the implant in native or regenerated bone, always in the antral area
  Other Names: ISQ

SUMMARY:
Compare ISQ values of implants placed in antral area in native bone vs regenerated bone with a follow-up at 3 months to compare values changes.

DETAILED DESCRIPTION:
The stability of dental implants is influenced by the type of bone in which the implant is placed. Native bone tends to provide better initial stability due to its density and quality, while regenerated bone, it is logical to think that it may present less stability due to the quality of the generated bone and the presence of defects in the treated area.

In this study it has been observed that after 3 months more stability is observed in the antral area, measured in ISQ resonance frequency in implants on regenerated bone, which surprises us and this result is explained in detail in said study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Total superior edentulism or antral zone edentulism
* Accepted study and signed inform consent

Exclusion Criteria:

* Patients under 23 years old
* Non accepted study or signed inform consent

Ages: 23 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group is made up of adult patients from the UEM Dental University Clinic, from September 2017 to September 2018, who attended the Master's Degree in Advanced Oral Implantology and who were informed of the study and signed the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Resonance frequency analysis (ISQ) measurements | 3 months
  The day of surgery, data were collected by vestibular and palatal, in addition, the mean of both measurements was taken and ISQ data were collected vertically to complete all the information. After 3 months of implant placement we recorded the same measurements and compared them in native and regenerated bone.

SECONDARY OUTCOMES:
Insertion torque measurements | During implant placement
  Analysis of the insertion torque values measured in Newtons per centimeter (Ncm) and comparing the results of both groups.
Changes in the marginal bone | 3 months
  Analysis of the changes in the marginal bone three months after implant placement

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Trapote Mateo, PhD, Study Director — European University of Madrid
Locations (1):
- Dental Clinic of the UEM, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No